CLINICAL TRIAL: NCT04603586
Title: A Prospective Phase Ⅱ Clinical Study of Stereotactic Radiotherapy Combined With Chemotherapy With Different Biological Effective Doses (<70gy vs. >70Gy) in Locally Advanced Pancreatic Cancer
Brief Title: Stereotactic Radiotherapy in Locally Advanced Pancreatic Cancer With Different Biological Effective Doses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhang Huo Jun, Director, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Changhai Hospit
Record Dates: First submitted 2020-10-15; First posted 2020-10-27 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Treatment
Keywords: SBRT; Locally Advanced Pancreatic Cancer; Biological Effective Dose
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): SBRT of BED<70Gy combined with Gemcitabine + albumin-bound paclitaxel
  Interventions: Radiation: SBRT; Drug: Chemotherapy
- Arm B (Experimental): SBRT of BED >70Gy combined with Gemcitabine + albumin-bound paclitaxel
  Interventions: Radiation: SBRT; Drug: Chemotherapy

INTERVENTIONS:
Radiation: SBRT — SBRT: in 5-6 fractions with CyberKnife
Drug: Chemotherapy — Gemcitabine 1000mg/m^2 and nab-paclitaxel 125mg/m^2, administered intravenously, on day 1 and 8 of a 21-day cycle for six cycles

SUMMARY:
The aim of this study is to compare the safety and efficacy of SBRT in LAPC with different biological effective dose (BED) (<70Gy Vs.>70Gy ) , to identify a dose range that could achieve better survival benefit and minimize the toxicity of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically verified pancreatic adenocarcinoma
* Imaging examinations confirmed locally advanced pancreatic cancer
* No previous radiotherapy, chemotherapy, immunotherapy or targeted therapy
* ECOG of 0 to1
* Age of 18 years or older
* Adequate bone marrow function, defined as: Absolute neutrophil count (ANC) ≥ 1.5×10^9 cells/L, leukocyte count≥ 3.5×10^9 cells/L, platelets ≥ 70×10^9 cells/L, hemoglobin ≥ 8.0 g/dl
* Adequate liver and renal, defined as: Albumin > 2.5 g/dL, total bilirubin < 3 mg/dL, creatinine < 2.0 mg/dL, AST<2.5 × ULN (Upper Limit of Normal) (0-64U/L), ALT<2.5 × ULN (0-64U/L)
* Adequate blood clotting function, defined as: international normalized ratio (INR) < 2 (0.9-1.1)
* Ability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Previously receiving radiotherapy, immunotherapy or targeted therapy
* Evidences of metastatic disease confirmed by chest CT or PET-CT
* ECOG ≥2
* Age <18 years
* Secondary malignancy
* Abnormal results of blood routine examinations and liver and kidney and coagulation tests
* Patients with active inflammatory bowel diseases or peptic ulcer
* Gastrointestinal bleeding or perforation within 6 months
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Medical history of symptomatic congestive heart failure: New York Heart Association Class III to IV
* Medical history of respiratory insufficiency
* Women who are pregnant or breastfeeding
* Participation in another clinical treatment trial
* Inability of the research subject or authorized legal representative to understand and the willingness to sign a written informed consent document

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Changhai hospital, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye Y, Zhu X, Zhao X, Jiang L, Cao Y, Zhang H. Biologically effective doses of 60-70Gy versus >70Gy of stereotactic body radiotherapy (SBRT) combined with chemotherapy in locally advanced pancreatic cancer: protocol of a single-centre, phase II clinical trial. BMJ Open. 2022 Aug 29;12(8):e049382. doi: 10.1136/bmjopen-2021-049382. PMID 36038164

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 60 | 59
Completed | 60 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 33 | 32 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 33 | 31 | 64
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Baseline characteristics [Count of Participants; unit: Participants] | 60 | 59 | 119

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free-Survival
Description: Progression-Free-Survival
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 60 | 59
month | 8.6 [7.5 to 9.6] | 11.3 [10.1 to 12.5]

2. Secondary Outcome: Adverse Events
Description: Adverse events
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 60 | 59
Participants | 58 | 57

3. Secondary Outcome: Overall Survival
Description: Overall Survival
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 60 | 59
months | 12.2 [10.9 to 13.5] | 17.2 [15.4 to 19.0]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 60/60 | 55/59
Serious Adverse Events (participants affected / at risk) | 26/60 | 25/59
Other Adverse Events (participants affected / at risk) | 58/60 | 57/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=60) | Arm B (N=59)
Leukopenia (Blood and lymphatic system disorders) | 11 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 9
Anemia (Blood and lymphatic system disorders) | 2 | 7
Nausea or vomiting (Gastrointestinal disorders) | 8 | 9
Fatigue (General disorders) | 7 | 8
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 8 | 5
Elevated alanine aminotransferase (Hepatobiliary disorders) | 4 | 8
Peripheral neurotoxicity (Nervous system disorders) | 6 | 7
Diarrhea (Gastrointestinal disorders) | 3 | 6
Fever (Infections and infestations) | 1 | 0
Blood bilirubin increased (Hepatobiliary disorders) | 0 | 1
Decreased appetite (Gastrointestinal disorders) | 14 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 4
Weight decreased (Metabolism and nutrition disorders) | 11 | 8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (N=60) | Arm B (N=59)
Leukopenia (Blood and lymphatic system disorders) | 49 | 50
Thrombocytopenia (Blood and lymphatic system disorders) | 41 | 39
Anemia (Blood and lymphatic system disorders) | 16 | 20
Nausea or vomiting (Gastrointestinal disorders) | 38 | 40
Fatigue (General disorders) | 51 | 48
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 35 | 41
Elevated alanine aminotransferase (Hepatobiliary disorders) | 37 | 42
Peripheral neurotoxicity (Nervous system disorders) | 11 | 10
Diarrhea (Gastrointestinal disorders) | 13 | 12
Fever (Infections and infestations) | 7 | 5
Blood bilirubin increased (Hepatobiliary disorders) | 3 | 4
Decreased appetite (Gastrointestinal disorders) | 48 | 51
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 | 22
Weight decreased (Metabolism and nutrition disorders) | 40 | 46
Constipation (Gastrointestinal disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Alopecia (General disorders) | 51 | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/86/NCT04603586/Prot_SAP_000.pdf